CLINICAL TRIAL: NCT05298735
Title: Pancreatic Calcium Handling in Islet Beta Cells in Patients With Type 1 Diabetes Mellitus
Acronym: Pancreas MEMRI
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC20142
Record Dates: First submitted 2022-03-10; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: Healthy volunteers with no known significant medical conditions
- Patients with type 1 diabetes: Patients with a diagnosis of type 1 diabetes (with or without detectable C-peptide)

SUMMARY:
Approximately 400,000 people are living with type 1 diabetes mellitus (T1DM) in the United Kingdom: one of the highest rates in the world. It is characterised by autoimmune loss of pancreatic beta cell mass leading to metabolic dysregulation, requiring lifelong insulin therapy. It is now recognised that there are micro-secretors of insulin and that preservation of insulin secretion in these cases is associated with decreased complications. Therefore, recent research has focussed on using immunomodulation to preserve pancreatic beta cell mass. Evaluation of novel therapies for T1DM requires reliable methods to measure beta-cell function, which is unattainable using traditional non-invasive imaging techniques. A new approach is manganese-enhanced magnetic resonance imaging (MEMRI). This proof-of-concept study was designed to investigate whether MEMRI can be used as a measure of beta-cell function in people with T1DM.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* No regular medications
* No known significant medical conditions

Exclusion Criteria:

* Inability to consent
* Renal failure (eGFR <30 mL/min/1.73 m2)
* Standard MRI contraindications
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 diabetes mellitus (with or without detectable C-peptide levels)
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Pancreatic calcium-handling: Rate of change of pancreatic T1 values with manganese-enhanced magnetic resonance imaging | 30 minutes after contrast administration

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided